CLINICAL TRIAL: NCT02203591
Title: Assessment of the Antimicrobial Efficacy of 3M CHG/IPA Preoperative Skin Preparation Against Resident Human Skin Flora on the Abdominal and Inguinal Regions
Brief Title: In Vivo Efficacy Study of Patient Preoperative Preps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EM-013260
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Bacterial Reduction Post-product Application
Keywords: surgical skin prep; CHG; IPA
MeSH Terms: interventions — chlorhexidine gluconate; 2-Propanol; Ethanol; Chromogranins; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- 3M CHG/IPA Prep C (Experimental): Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Prep C
- 3M CHG/IPA Prep CH (Experimental): Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Prep CH
- ChloraPrep (Active Comparator): Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: ChloraPrep
- Normal Saline (Placebo Comparator): Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: 3M CHG/IPA Prep C — Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Other Names: Chlorhexidine Gluconate and Isopropyl Alcohol; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%; CHG 2%/IPA 70%
  Arms: 3M CHG/IPA Prep C
Drug: 3M CHG/IPA Prep CH — Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Other Names: Chlorhexidine Gluconate and Isopropyl Alcohol; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%; CHG 2%/IPA 70%
  Arms: 3M CHG/IPA Prep CH
Drug: ChloraPrep — Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Other Names: ChloraPrep Patient Preoperative Skin Preparation; ChloraPrep One-Step; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%; CHG2%/IPA 70%; Chlorhexidine Gluconate and Isopropyl Alcohol
  Arms: ChloraPrep
Drug: Normal Saline — Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Other Names: Sodium Chloride 0.9%; Saline
  Arms: Normal Saline

SUMMARY:
The objective of this study is to demonstrate the antimicrobial efficacy of the 3M CHG/IPA Prep on skin flora of the abdominal and inguinal regions of human subjects.

DETAILED DESCRIPTION:
The primary efficacy is evaluated by demonstration that the product provides a lower bound of the 95% confidence interval of percent responders that is greater than or equal to 70% On the abdominal site, a responder is defined as a subject with a 2-log10/cm2 bacterial reduction at 10 minutes and for whom the skin flora does not return to baseline at 6 hours.

On the inguinal site, a responder is defined as a subject with a 3-log10/cm2 bacterial reduction at 10 minutes and for whom the skin flora does not return to baseline at 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race
* Subjects in good health
* Minimum skin flora baseline requirements on abdomen and groin

Exclusion Criteria:

* Any tattoos, scars, breaks in the skin, or any form of dermatitis, or other skin disorders (including acne) on the applicable test area
* Topical antimicrobial exposure within 14 days prior to screening and treatment days
* Use of systemic or topical antibiotics, steroid medications, or any other products known to affect the normal microbial flora of the skin within 14 days prior to screening and treatment days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Miller, ADN, Principal Investigator — Independent Consultant
Locations (1):
- BioScience Laboratories, Inc., Bozeman, Montana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomized, paired comparison design where each subject received 2 of the planned treatments, 1 on the left side & 1 on the right. Each subject provided 2 abdomen test sties, left & right and/or 2 inguen test sites, left & right.
  569 subjects were randomized for the abdomen region & 404 subjects randomized for the inguen region resulting in 738 subjects providing 1946 applications of test products on 2 anatomical regions.
Units Other Than Participants: test sites on skin
Groups:
- 3M CHG/IPA Prep C - Abdominal; 3M CHG/IPA Prep CH - Abdominal; ChloraPrep - Abdominal; Normal Saline - Abdominal: Applied topically to the abdominal region for 30 seconds.
- 3M CHG/IPA Prep C - Inguinal; 3M CHG/IPA Prep CH - Inguinal; ChloraPrep - Inguinal; Normal Saline - Inguinal: Applied topically to the inguinal region for 2 minutes.
Period: Overall Study
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Started | 343; 343 test sites on skin | 344; 344 test sites on skin | 347; 347 test sites on skin | 104; 104 test sites on skin | 242; 242 test sites on skin | 244; 244 test sites on skin | 248; 248 test sites on skin | 74; 74 test sites on skin
Completed | 196; 196 test sites on skin | 202; 202 test sites on skin | 196; 196 test sites on skin | 59; 59 test sites on skin | 208; 208 test sites on skin | 209; 209 test sites on skin | 219; 219 test sites on skin | 61; 61 test sites on skin
Not Completed | 147; 147 test sites on skin | 142; 142 test sites on skin | 151; 151 test sites on skin | 45; 45 test sites on skin | 34; 34 test sites on skin | 35; 35 test sites on skin | 29; 29 test sites on skin | 13; 13 test sites on skin
Not completed — Did not meet treatment day baseline | 147 | 141 | 150 | 45 | 33 | 35 | 29 | 12
Not completed — Discontinued early due to compromised test sites | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects with average screening day baseline counts of greater than or equal to 3.00 log10 CFU/cm2 bilaterally on the abdominal region and/or greater than or equal to 5.00 log10 CFU/cm2 bilaterally on the inguinal region were included in the analysis.
Units Other Than Participants: test sites on skin
Groups:
- 3M CHG/IPA Prep C - Abdominal; 3M CHG/IPA Prep CH - Abdominal; ChloraPrep - Abdominal; Saline - Abdominal: Applied topically for 30 seconds to the abdominal test site
- 3M CHG/IPA Prep C - Inguinal; 3M CHG/IPA Prep CH - Inguinal; ChloraPrep - Inguinal; Saline - Inguinal: Applied topically for 2 minutes to the inguinal test site
- Total: Total of all reporting groups
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Saline - Inguinal | Total
Number analyzed (Participants) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74 | 1946
Number analyzed (test sites on skin) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74 | 1946
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 333 | 338 | 332 | 102 | 236 | 236 | 245 | 73 | 1895
  >=65 years | 10 | 6 | 15 | 2 | 6 | 8 | 3 | 1 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 99 | 105 | 32 | 56 | 64 | 67 | 23 | 538
  Male | 251 | 245 | 242 | 72 | 186 | 180 | 181 | 51 | 1408
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 6 | 3 | 2 | 3 | 4 | 5 | 0 | 28
  Asian | 8 | 8 | 9 | 1 | 5 | 8 | 7 | 2 | 48
  Black or African American | 6 | 2 | 7 | 1 | 1 | 1 | 0 | 0 | 18
  Hispanic / Latino | 13 | 9 | 15 | 5 | 9 | 11 | 14 | 0 | 76
  Native Hawaiin or Other Pacific Islander | 3 | 2 | 1 | 0 | 2 | 0 | 2 | 0 | 10
  White | 308 | 320 | 316 | 96 | 222 | 222 | 221 | 71 | 1776
  Other | 7 | 3 | 3 | 1 | 2 | 4 | 6 | 2 | 28
Region of Enrollment [Number; unit: participants]
  United States | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74 | 973

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate
Description: On the abdominal region a responder is a subject with a 2 log10/cm^2 bacterial reduction at 10 minutes and for whom the skin flora does not return to baseline at the 6-hour sample collection time.
  On the inguinal region a responder is a subject with a 3 log10/cm^2 bacterial reduction at 10 minutes and for whom the skin flora does not return to baseline at the 6-hour sample collection time.
Time Frame: baseline, 10 minutes post-product application and 6 hours post-product application
Measure: Count of Participants; unit: Participants
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 196 | 202 | 196 | 59 | 208 | 209 | 219 | 61
Participants | 159 | 165 | 163 | 5 | 81 | 98 | 116 | 1
Statistical Analysis 1: Comparison: 3M CHG/IPA Prep C - Abdominal vs Normal Saline - Abdominal; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: 3M CHG/IPA Prep CH - Abdominal vs Normal Saline - Abdominal; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: ChloraPrep - Abdominal vs Normal Saline - Abdominal; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: 3M CHG/IPA Prep C - Inguinal vs Normal Saline - Inguinal; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 5: Comparison: 3M CHG/IPA Prep CH - Inguinal vs Normal Saline - Inguinal; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 6: Comparison: ChloraPrep - Inguinal vs Normal Saline - Inguinal; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 7: Comparison: 3M CHG/IPA Prep C - Abdominal; Test type: Other — 95% confidence interval generation; Mean value = 81.1, 95% CI 2-sided [75.6 to 86.6]
Statistical Analysis 8: Comparison: 3M CHG/IPA Prep CH - Abdominal; Test type: Other — 95% confidence interval generation; Mean value = 81.7, 95% CI 2-sided [76.3 to 87.1]
Statistical Analysis 9: Comparison: ChloraPrep - Abdominal; Test type: Other — 95% confidence interval generation; Mean value = 83.2, 95% CI 2-sided [77.9 to 88.4]
Statistical Analysis 10: Comparison: 3M CHG/IPA Prep C - Inguinal; Test type: Other — 95% confidence interval generation; Mean value = 38.9, 95% CI 2-sided [32.3 to 45.6]
Statistical Analysis 11: Comparison: 3M CHG/IPA Prep CH - Inguinal; Test type: Other — 95% confidence interval generation; Mean value = 46.9, 95% CI 2-sided [40.1 to 53.7]
Statistical Analysis 12: Comparison: ChloraPrep - Inguinal; Test type: Other — 95% confidence interval generation; Mean value = 53.0, 95% CI 2-sided [46.3 to 59.6]

2. Primary Outcome: Alternative Primary
Description: 10 minute log reduction
Time Frame: Baseline and 10 minutes
Measure: Mean (Standard Deviation); unit: log10/cm^2
Arm/Group | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal
Number analyzed (Participants) | 208 | 209 | 219
log10/cm^2 | 2.84 (1.19) | 2.99 (1.12) | 3.17 (1.24)
Statistical Analysis 1: Comparison: 3M CHG/IPA Prep C - Inguinal vs ChloraPrep - Inguinal; Test type: Non-Inferiority — A non-inferior margin of 0.5 log10/cm^2; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.57 to -0.10], Standard Error of Mean 0.12 — 3M CHG/IPA C - Inguinal minus ChloraPrep - Inguinal
Statistical Analysis 2: Comparison: 3M CHG/IPA Prep CH - Inguinal vs ChloraPrep - Inguinal; Since there are two investigational products a Hochberg step-up procedure was used to adjust for multiplicity; Test type: Non-Inferiority — A non-inferior margin of 0.5 log10/cm^2; Mean Difference (Final Values) = -0.18, 97.5% CI 2-sided [-0.44 to 0.74], Standard Error of Mean 0.11 — 3M CHG/IPA CH - Inguinal minus ChloraPrep - Inguinal

3. Secondary Outcome: Reduction of Skin Flora 6 Hours Post-treatment
Description: Log10/cm^2 reduction of skin flora, relative to treatment day baseline, 6 hours post-treatment application
Time Frame: 6 hours
Population: The primary analysis dataset used a mITT population. Subjects were excluded who did not meet the treatment day baseline requirements (stated in the Inclusion/Exclusion criteria).
Measure: Mean (Standard Deviation); unit: log10/cm^2 skin flora
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 196 | 202 | 196 | 59 | 208 | 209 | 219 | 61
log10/cm^2 skin flora | 2.83 (0.851) | 2.86 (0.899) | 2.83 (0.971) | 1.00 (0.971) | 3.46 (1.312) | 3.49 (1.329) | 3.69 (1.286) | 1.23 (0.732)
Statistical Analysis 1: Comparison: 3M CHG/IPA Prep C - Abdominal; Test type: Other — Calculate mean value; Mean value = 2.83, Standard Deviation 0.85
Statistical Analysis 2: Comparison: 3M CHG/IPA Prep CH - Abdominal; Test type: Other — Calculate mean value; Mean value = 2.86, Standard Deviation 0.90
Statistical Analysis 3: Comparison: ChloraPrep - Abdominal; Test type: Other — Calculate mean value; Mean value = 2.83, Standard Deviation 0.97
Statistical Analysis 4: Comparison: Normal Saline - Abdominal; Test type: Other — Calculate mean value; Mean value = 1.00, Standard Deviation 0.97
Statistical Analysis 5: Comparison: 3M CHG/IPA Prep C - Inguinal; Test type: Other — Calculate mean value; Mean value = 3.46, Standard Deviation 1.31
Statistical Analysis 6: Comparison: 3M CHG/IPA Prep CH - Inguinal; Test type: Other — Calculate mean value; Mean value = 3.49, Standard Deviation 1.33
Statistical Analysis 7: Comparison: ChloraPrep - Inguinal; Test type: Other — Calculate mean value; Mean value = 3.69, Standard Deviation 1.29
Statistical Analysis 8: Comparison: Normal Saline - Inguinal; Test type: Other — Calculate mean value; Mean value = 1.23, Standard Deviation 0.73

4. Secondary Outcome: Reduction of Skin Flora 10 Minutes Post-treatment
Description: Log10/cm^2 reduction of skin flora, relative to treatment day baseline (log10/cm^2) at 10 minutes post-treatment application
Time Frame: 10 minutes
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10/cm^2 skin flora
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 196 | 202 | 196 | 59 | 208 | 209 | 219 | 61
log10/cm^2 skin flora | 2.78 (0.935) | 2.73 (1.002) | 2.75 (0.973) | 0.76 (0.814) | 2.84 (1.191) | 2.99 (1.125) | 3.17 (1.243) | 1.01 (0.668)
Statistical Analysis 1: Comparison: 3M CHG/IPA Prep C - Abdominal; Test type: Other — Calculate mean value; Mean value = 2.78, Standard Deviation 0.94
Statistical Analysis 2: Comparison: 3M CHG/IPA Prep CH - Abdominal; Test type: Other — Calculate mean value; Mean value = 2.73, Standard Deviation 1.00
Statistical Analysis 3: Comparison: ChloraPrep - Abdominal; Test type: Other — Calculate mean value; Mean value = 2.75, Standard Deviation 0.97
Statistical Analysis 4: Comparison: Normal Saline - Abdominal; Test type: Other — Calculate mean value; Mean value = 0.76, Standard Deviation 0.81
Statistical Analysis 5: Comparison: 3M CHG/IPA Prep C - Inguinal; Test type: Other — Calculate mean value; Mean value = 2.84, Standard Deviation 1.19
Statistical Analysis 6: Comparison: 3M CHG/IPA Prep CH - Inguinal; Test type: Other — Calculate mean value; Mean value = 2.99, Standard Deviation 1.12
Statistical Analysis 7: Comparison: ChloraPrep - Inguinal; Test type: Other — Calculate mean value; Mean value = 3.17, Standard Deviation 1.24
Statistical Analysis 8: Comparison: Normal Saline - Inguinal; Test type: Other — Calculate mean value; Mean value = 1.01, Standard Deviation 0.67

5. Secondary Outcome: Skin Flora Recovery 6-hours Post-treatment
Description: Log10/cm^2 recovery of skin flora at 6 hours following application of treatment
Time Frame: 6 hours post-treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10/cm^2 skin flora
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 196 | 201 | 196 | 59 | 208 | 209 | 219 | 60
log10/cm^2 skin flora | 0.80 (0.840) | 0.74 (0.789) | 0.81 (0.935) | 2.65 (0.886) | 2.76 (1.202) | 2.73 (1.220) | 2.58 (1.182) | 4.85 (0.749)
Statistical Analysis 1: Comparison: 3M CHG/IPA Prep C - Abdominal; Test type: Other — Calculate mean value; Mean value = 0.80, Standard Deviation 0.84
Statistical Analysis 2: Comparison: 3M CHG/IPA Prep CH - Abdominal; Test type: Other — Calculate mean value; Mean value = 0.74, Standard Deviation 0.79
Statistical Analysis 3: Comparison: ChloraPrep - Abdominal; Test type: Other — Calculate mean value; Mean value = 0.81, Standard Deviation 0.94
Statistical Analysis 4: Comparison: Normal Saline - Abdominal; Test type: Other — Calculate mean value; Mean value = 2.65, Standard Deviation 0.89
Statistical Analysis 5: Comparison: 3M CHG/IPA Prep C - Inguinal; Test type: Other — Calculate mean value; Mean value = 2.76, Standard Deviation 1.20
Statistical Analysis 6: Comparison: 3M CHG/IPA Prep CH - Inguinal; Test type: Other — Calculate mean value; Mean value = 2.73, Standard Deviation 1.22
Statistical Analysis 7: Comparison: ChloraPrep - Inguinal; Test type: Other — Calculate mean value; Mean value = 2.58, Standard Deviation 1.18
Statistical Analysis 8: Comparison: Normal Saline - Inguinal; Test type: Other — Calculate mean value; Mean value = 4.85, Standard Deviation 0.75

6. Secondary Outcome: Skin Flora Recovery 10 Minutes Post-treatment
Description: Log10/cm^2 recovery of skin flora at 10 minutes following application of study treatments.
Time Frame: 10 minute post-product application
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10/cm^2 skin flora
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 196 | 201 | 196 | 59 | 208 | 208 | 218 | 60
log10/cm^2 skin flora | 0.85 (0.947) | 0.88 (0.984) | 0.90 (0.938) | 2.88 (0.703) | 3.39 (1.096) | 3.21 (1.042) | 3.08 (1.137) | 5.08 (0.676)
Statistical Analysis 1: Comparison: 3M CHG/IPA Prep C - Abdominal; Test type: Other — Calculate mean value; Mean value = 0.85, Standard Deviation 0.95
Statistical Analysis 2: Comparison: 3M CHG/IPA Prep CH - Abdominal; Test type: Other — Calculate mean value; Mean value = 0.87, Standard Deviation 0.98
Statistical Analysis 3: Comparison: ChloraPrep - Abdominal; Test type: Other — Calculate mean value; Mean value = 0.89, Standard Deviation 0.94
Statistical Analysis 4: Comparison: Normal Saline - Abdominal; Test type: Other — Calculate mean value; Mean value = 2.88, Standard Deviation 0.70
Statistical Analysis 5: Comparison: 3M CHG/IPA Prep C - Inguinal; Test type: Other — Calculate mean value; Mean value = 3.39, Standard Deviation 1.10
Statistical Analysis 6: Comparison: 3M CHG/IPA Prep CH - Inguinal; Test type: Other — Calculate mean value; Mean value = 3.21, Standard Deviation 1.04
Statistical Analysis 7: Comparison: ChloraPrep - Inguinal; Test type: Other — Calculate mean value; Mean value = 3.08, Standard Deviation 1.14
Statistical Analysis 8: Comparison: Normal Saline - Inguinal; Test type: Other — Calculate mean value; Mean value = 5.08, Standard Deviation 0.68

7. Secondary Outcome: Skin Flora Baseline for the Abdomen and Inguinal Region.
Description: Log10/cm^2 baseline skin flora for abdominal and inguinal regions
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10/cm^2 skin flora
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 196 | 202 | 196 | 59 | 208 | 209 | 219 | 61
log10/cm^2 skin flora | 3.63 (0.460) | 3.61 (0.479) | 3.64 (0.487) | 3.64 (0.533) | 6.23 (0.604) | 6.21 (0.563) | 6.27 (0.618) | 6.09 (0.626)
Statistical Analysis 1: Comparison: 3M CHG/IPA Prep C - Abdominal; Test type: Other — Calculate mean value; Mean value = 3.63, Standard Deviation 0.46
Statistical Analysis 2: Comparison: 3M CHG/IPA Prep CH - Abdominal; Test type: Other — Calculate mean value; Mean value = 3.61, Standard Deviation 0.48
Statistical Analysis 3: Comparison: ChloraPrep - Abdominal; Test type: Other — Calculate mean value; Mean value = 3.64, Standard Deviation 0.49
Statistical Analysis 4: Comparison: Normal Saline - Abdominal; Test type: Other — Calculate mean value; Mean value = 3.64, Standard Deviation 0.53
Statistical Analysis 5: Comparison: 3M CHG/IPA Prep C - Inguinal; Test type: Other — Calculate mean value; Mean value = 6.23, Standard Deviation 0.60
Statistical Analysis 6: Comparison: 3M CHG/IPA Prep CH - Inguinal; Test type: Other — Calculate mean value; Mean value = 6.22, Standard Deviation 0.56
Statistical Analysis 7: Comparison: ChloraPrep - Inguinal; Test type: Other — Calculate mean value; Mean value = 6.27, Standard Deviation 0.62
Statistical Analysis 8: Comparison: Normal Saline - Inguinal; Test type: Other — Calculate mean value; Mean value = 6.09, Standard Deviation 0.63

8. Secondary Outcome: Safety as Assessed by Skin Irritation (Dryness, Edema, Erythema, Rash) Rating Score
Description: Skin irritation (dryness, edema, erythema, rash) assessed on the test sites using a 0-3 rating scale; 0 = no reaction, 1 = mild, 2 = moderate, 3 = severe.
Time Frame: Baseline
Population: The primary safety analysis data set used an Intent-To-Treat (ITT) population
Measure: Number; unit: participants
Units Other Than Participants: test sites on skin
Groups:
- 3M CHG/IPA Prep C - Abdominal: Applied topically to the abdominal region for 30 seconds.
  .
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74
Number analyzed (test sites on skin) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74
participants
  Dryness-No Reaction (0) | 343 | 344 | 347 | 104 | 240 | 244 | 248 | 74
  Dryness-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dryness-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-No Reaction (0) | 343 | 344 | 347 | 104 | 240 | 244 | 248 | 74
  Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-No Reaction (0) | 340 | 343 | 347 | 104 | 239 | 243 | 247 | 74
  Erythema-Mild (1) | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 0
  Erythema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-No Reaction (0) | 343 | 344 | 347 | 104 | 240 | 244 | 248 | 74
  Rash-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Safety Assessed as Skin Irritation (Dryness, Edema, Erythema, Rash) Rating Score
Description: Skin irritation (dryness, edema, erythema, rash) assessed on the test sites using a 0-3 rating scale; 0=no reaction, 1=mild, 2=moderate, 3=severe
Time Frame: 10 minutes post-treatment
Population: The primary safety analysis data set used an Intent to Treat population
Measure: Number; unit: participants
Units Other Than Participants: test sites on skin
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74
Number analyzed (test sites on skin) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74
participants
  Dryness-No Reaction (0) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 73
  Dryness-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Dryness-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-No Reaction | 343 | 344 | 347 | 104 | 242 | 244 | 247 | 74
  Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-No Reaction (0) | 341 | 343 | 345 | 104 | 240 | 242 | 243 | 73
  Erythema-Mild (1) | 2 | 1 | 2 | 0 | 2 | 2 | 5 | 1
  Erythema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-No Reaction (0) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74
  Rash-Mild(1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Safety as Assessed by Skin Irritation Score
Description: Skin irritation rating (0-3) scores for dryness, edema, erythema and rash; 0 = no reaction, 1 = mild, 2 = moderate, 3 = severe.
Time Frame: 6 hours post-treatment
Population: The primary safety analysis dataset used an Intent-To-Treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74
Participants
  Dryness-No Reaction (0) | 334 | 330 | 336 | 101 | 240 | 240 | 241 | 73
  Dryness-Mild (1) | 9 | 14 | 10 | 3 | 2 | 4 | 7 | 1
  Dryness-Moderate (2) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-No Reaction (0) | 343 | 344 | 347 | 104 | 242 | 244 | 248 | 74
  Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-No Reaction (0) | 310 | 310 | 332 | 98 | 227 | 220 | 236 | 72
  Erythema-Mild (1) | 32 | 33 | 15 | 6 | 15 | 24 | 12 | 2
  Erythema-Moderate (2) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-No Reaction (0) | 339 | 337 | 342 | 103 | 230 | 231 | 229 | 66
  Rash-Mild (1) | 4 | 7 | 5 | 1 | 12 | 13 | 19 | 8
  Rash-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected after treatment; by definition, all AEs were treatment-emergent.
Arm/Group | 3M CHG/IPA Prep C - Abdominal | 3M CHG/IPA Prep CH - Abdominal | ChloraPrep - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep C - Inguinal | 3M CHG/IPA Prep CH - Inguinal | ChloraPrep - Inguinal | Normal Saline - Inguinal
All-Cause Mortality (participants affected / at risk) | 0/343 | 0/344 | 0/347 | 0/104 | 0/242 | 0/244 | 0/248 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/343 | 0/344 | 0/347 | 0/104 | 0/242 | 0/244 | 0/248 | 0/74
Other Adverse Events (participants affected / at risk) | 2/343 | 3/344 | 1/347 | 0/104 | 2/242 | 3/244 | 0/248 | 0/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3M CHG/IPA Prep C - Abdominal (N=343) | 3M CHG/IPA Prep CH - Abdominal (N=344) | ChloraPrep - Abdominal (N=347) | Normal Saline - Abdominal (N=104) | 3M CHG/IPA Prep C - Inguinal (N=242) | 3M CHG/IPA Prep CH - Inguinal (N=244) | ChloraPrep - Inguinal (N=248) | Normal Saline - Inguinal (N=74)
Mild severity (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 0
Moderate severity (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not related to product (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Possibly related to products (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Probably related to product (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 1 | 2 | 0 | 0
Anticipated (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 2 | 3 | 0 | 0
Unexpected (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes